CLINICAL TRIAL: NCT07058896
Title: Unravelling The Optimisation And Consolidation Of Motor Skills In People With Multiple Sclerosis With Severe Gait Impairment Via High Intensity Task Oriented Circuit Training: A Feasibility Study
Brief Title: Unravelling The Optimisation And Consolidation Of Motor Skills In People With Multiple Sclerosis With Severe Gait Impairment: A Feasibility Study
Acronym: UNLOCK MS SGI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, MD, PhD, University Hospital of Ferrara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNLOCK_MS_SGI_HITOCT
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; high intensity training; motor learning; circuit training; rehabilitation; balance; mobility
MeSH Terms: conditions — Multiple Sclerosis | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- High Intensity Task Oriented Circuit Training + Telerehabilitation (Experimental): Participants will receive 12 sessions of high-intensity, task-focused circuit training, three times a week for four weeks. Each 180-minute session includes 108 minutes of active training, with three rounds of exercises at different stations. Activities will focus on motor skills like standing, walking, transfers, and wheelchair use. If walking isn't possible, upper limb training will be included instead.
  After hospital treatment, participants will continue with 36 asynchronous telerehabilitation sessions over 12 weeks, including monthly televisits, using low-cost, commercially available technology.
  Interventions: Behavioral: High intensity task oriented circuit training + Telerehabilitation

INTERVENTIONS:
Behavioral: High intensity task oriented circuit training + Telerehabilitation — Participants will receive 12 sessions of high-intensity, task-oriented circuit training, three times a week for four weeks. Each session will last 180 minutes, with 108 minutes of active training. Each session will include three rounds, each lasting 51 minutes. During each round, participants will rotate between stations working for six minutes at each station, followed by three minutes of rest. The stations will focus on key motor skills, including sit-to-stand transitions, walking, standing, bed mobility and transfers, stepping, and wheelchair use. If participants are unable to walk, the walking station will be replaced by upper limb function station.
  After in-hospital treatment participants will receive 36 sessions of asynchronous telerehabilitation, three times a week for 12 weeks. Including monthly televisits with the physiotherapist. This intervention will be supported by low-cost, off-the-shelf technology for treatment delivery and monitoring.

SUMMARY:
Multiple sclerosis (MS) is a progressive neurological disorder that often leads to severe gait impairment, limiting mobility and reducing the patient's quality of life. Motor rehabilitation has shown positive effects in people with MS (PwMS), but its efficacy tends to decrease as disability severity increases. High-intensity, task-oriented circuit training based on the principles of motor learning has been proposed as a potential strategy to improve motor function in severely impaired individuals.

This approach combines the benefits of high-intensity training to the motor learning principles to enhance motor skills improvement and retention.

The main questions it aims to answer are:

* Can high-intensity, task oriented training in PwMS with severe gait impairment be feasible, safe and effective in enhancing motor function?
* Can telerehabilitation maintain the benefits in gait and balance gained via circuit training for a six month period?

Participants will:

* Complete 12 session ( three hour each, three times a week) of high-intensity task oriented circuit training administered in a hospital setting. The training will target key motor skills such as walking, stepping, sit to stand, wheelchair, standing and bed mobillity.
* Engage in 3 months of asynchronous telerehabilitation (without physiotherapist supervision), including monthly televisits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary or secondary progressive multiple sclerosis according to the McDonald criteria.
* Mini-Mental State Examination (MMSE) score > 24.
* Expanded Disability Status Scale (EDSS) score ≥ 6.5.

Exclusion Criteria:

* Presence of other psychiatric or neurological disorders.
* Cardiopulmonary, renal, or liver diseases.
* Pregnancy.
* Modifications in drug treatment within the last 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Static Balance | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  The change in static balance will be assessed using the Berg Balance Scale

SECONDARY OUTCOMES:
Change in Walking capacity | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Walking capacity will be assessed through the 6 Minute Walking Test
Change in Walking speed | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Walking speed will be assesed through the Timed 25 Foot Walk
Change in mobility, balance, walking ability, and fall risk | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Mobility, balance, walking ability, and fall risk will be assessed through Timed Up and Go Test
Change in quantitative mobility and leg function performance | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Leg function performance and quantitative mobility assessed through Timed 25 Foot Walk
Change in auditory information processing speed and flexibility | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Paced Auditory Serial Addition Test will be used to assess auditory information processing speed and flexibility
Changes in functional lower extremity strength | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Five Times Sit to Stand will be used to assess functional lower extremity strength
Change in cardiovascular fitness | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Cardiovascular fitness will be assessed with 6 Minute Push Test
Change in Subjective Trait Fatigue | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Change in subjective trait fatigue will be assessed through Modified Fatigue Impact Scale
Change in impacts of multiple sclerosis in people' lifes | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  The impact of multiple sclerosis in people' lifes will be assessed through Multiple Sclerosis Impact Scale 29.
Change in balance confidence | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Change in balance confidence will be assessed through Activity-Specific Balance Confidence Scale.
Change in functional performance of the upper extremity | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Functional performance of the upper extremity will assessed through Action Research Arm Test
Change in self perceived manual ability | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  Self perceived manual ability will be assessed through ABILHAND 26
Change in Walking Fatigability | Baseline testing (T0), score changes after the 4 weeks in-hospital treatment (T1), score changes after the 3-months asynchronous telerehabilitation intervention (T1) and score changes at follow up, 3 months after telerehabilitation intervetion (T3)
  The Distance Walking Index will be used to assess the Change in Walking Fatigability

CONTACTS AND LOCATIONS:
Locations (1):
- Ferrara University Hospital, Ferrara, FE, Italy